CLINICAL TRIAL: NCT03284515
Title: Vaccination In Pregnancy Gene Signature: VIP Signature Study
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: Innovative Medicine Initiative (Unknown); Max Planck Institute for Infection Biology (Other)
Responsible Party: Sponsor
Other Study IDs: 17.0060
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Pregnancy Related; Vaccination
MeSH Terms: interventions — Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken from the women prior to and 24 hours following vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All women: Women who are between 16-32 weeks gestation and who have not previously received a pertussis vaccination in pregnancy.
  Interventions: Biological: Vaccination with a pertussis containing vaccine

INTERVENTIONS:
Biological: Vaccination with a pertussis containing vaccine — Vaccination with a pertussis containing vaccine

SUMMARY:
A study investigating gene expression profiles in pregnant women in response to a pertussis containing vaccination in pregnancy.

DETAILED DESCRIPTION:
Vaccinations are a vital part of ensuring population health, but there is a continued need for new and improved vaccines to be developed and this process of design and development can be both slow and expensive. Vaccination in pregnancy against pathogens such as pertussis, influenza and tetanus is a routine part of antenatal care in many countries. The principle behind this approach is that through vaccination the amount of disease specific antibody is increased in the woman and there is therefore an increase in transplacental transfer to the fetus providing protection for infants after birth. In the UK vaccination against pertussis is recommended from 16 weeks gestation and against influenza at any gestation within the influenza season. There is evidence that pertussis vaccination in pregnancy is highly effective against pertussis in infants too young to be protected by the routine infant immunisation programme (Amirthalingam G et al, 2014, Dabrera G et al, 2015). There is also evidence that this is a safe strategy in pregnancy to protect newborn infants (Donegan K et al, 2014) with no evidence of adverse clinical outcomes for mother or infant.

The BioVacSafe project has been designed to develop techniques which can be used to understand more about biomarkers of safety in individuals' response to vaccines. This will improve our understanding of how reactogenicity can be identified earlier, how adverse reactions can be identified and classified and how individuals interact with vaccines, specifically in conditions of health and disease. Since the start of the BioVacSafe project the importance of vaccination in pregnancy has become better understood and it has become important to include pregnant women as participants in this project. Pregnancy is a time of altered immunity and it may be that there are differences in gene signatures following vaccination in pregnant women compared with non-pregnant women. Insights into this could be extremely important in the development of new vaccines for this population.

Safety of vaccination in pregnancy is of primary importance to pregnant women and their partners, clinical trials investigators, ethics committees, vaccine manufacturers and regulators. Determining specific genetic signatures following vaccination may accelerate vaccine development by predicting possible adverse events early in the development process.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at a gestation of 16-32 weeks
* No contraindications to vaccination according to the green book
* No known immunodeficiency
* Able to understand the details of the study and willing to provide informed consent

Exclusion Criteria:

* Having received a pertussis containing vaccine within the last 12 months
* Contraindications to vaccination according to the green book

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women at between 16-32 weeks gestation who have not yet received the pertussis vaccination in pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Gene expression profiles | 24 hours
  Gene expression profiles in blood samples from pregnant women following vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Personal details of the participants will be collected to allow us to contact them if necessary. This information will be stored securely and will not leave St. George's, University of London. Some limited demographic and medical information may be shared with researchers at Imperial College London and the Max Planck Institute for Infection Biology both of which are part of this study and the wider BioVacSafe consortium.